CLINICAL TRIAL: NCT04481607
Title: A Phase I, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerance, Efficacy and Pharmacokinetics of TQB3454 Tablets
Brief Title: A Study to Evaluate the Tolerance, Efficacy and Pharmacokinetics of TQB3454 Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3454-I-02
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Advanced Solid Tumor or Hematologic Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3454 tablets (Experimental): TQB3454 tablets administered orally once. Then TQB3454 tablets administered orally, once daily in 28-day cycle after 7 days of first administration.
  Interventions: Drug: TQB3454

INTERVENTIONS:
Drug: TQB3454 — TQB3454 tablets is a small molecule oral drug.

SUMMARY:
This is a open-label, multicenter, phase I study to evaluate tolerance and pharmacokinetics of TQB3454 tablets in subjects with advanced solid tumor or hematologic tumor.

ELIGIBILITY:
Inclusion Criteria:

- 1. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1; Life expectancy ≥12 weeks.

2. Advanced solid tumors or hematological malignancy. 3. Adequate laboratory indicators. 4. No pregnant or breastfeeding women, and a negative pregnancy test. 5. Understood and Signed an informed consent form.

Exclusion Criteria:

* 1. Has central nervous system metastasis or system leukemia. 2.Previous anti-tumor treatment:

  1. Has received IDH1 mutation inhibitor.
  2. Has received systemic anti-tumor therapy or radiotherapy within 14 days before the first dose.
  3. Has received oral targeted drugs, less than 5 drug half-lives from first dose.
  4. The related toxicity of previous anti-tumor therapy has not recovered to CTCAE ≤ grade 2, except for hair loss.

     3.Complicated disease and medical history:

  <!-- -->

  1. Active hepatitis B or hepatitis C.
  2. Abnormal kidney.
  3. Abnormal cardiovascular and cerebrovascular.
  4. Abnormal gastrointestinal.
  5. Has medical history of immunodeficiency.
  6. Has bleeding (hemoptysis), coagulopathy, or been using warfarin, aspirin, and other antiplatelet agglutination drugs.
  7. Has uncontrollable systemic bacterial, fungal or viral active infections.
  8. Has medical history of idiopathic pulmonary fibrosis,or tissue pneumonia.
  9. Has allergic constitution or previous severe allergy; or known allergy to ingredients of study drug.
  10. Has neurological or mental disorders.
  11. Has a history of drug abuse or drug addict.
  12. Has received major surgery, open biopsy, or obvious traumatic injury within 4 weeks before the first dose.
  13. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

      4. Has participated in other clinical trials within 30 days before participating in this trial.

      5. Female patients during pregnancy or lactation. 6. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

      7. criteria for solid tumors:

  <!-- -->

  1. Has any signs of bleeding constitution.
  2. Has any CTCAE ≥ grade 3 bleeding or bleeding event,within 4 weeks before the first dose.
  3. Has unhealed wounds, fractures, active ulcers of the stomach and duodenum, ulcerative colitis and other digestive tract diseases.
  4. Imaging (CT or MRI) shows that the tumor has invaded the circumference of important blood vessels.
  5. Has uncontrollable pleural effusion, pericardial effusion or ascites that still need repeated drainage.

criteria for blood tumor:

a) Has severe life-threatening leukemia complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 28 days
  MTD was defined as the dose in which more than 2 of up to 6 patients developed a DLT.

SECONDARY OUTCOMES:
Cmax | Hour 0(pre-dose), 0.5, 1, 2, 3, 5, 8, 10, 24, 48, 72, 120, 168 hours post-dose on single dose;
  Cmax is the maximum plasma concentration of TQB3454 or metabolite(s).
Tmax | Hour 0(pre-dose), 0.5, 1, 2, 3, 5, 8, 10, 24, 48, 72, 120, 168 hours post-dose on single dose;
  To characterize the pharmacokinetics of TQB3454 by assessment of time to reach maximum plasma concentration.
AUC0-t | Hour 0(pre-dose), 0.5, 1, 2, 3, 5, 8, 10, 24, 48, 72, 120, 168 hours post-dose on single dose;
  To characterize the pharmacokinetics of TQB3454 by assessment of area under the plasma concentration time curve from zero to infinity.
Objective response rate (ORR) | up to 60 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).
Progression-free survival (PFS) | Up to 60 weeks
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
2-hydroxyglutaric acid | Hour 0(pre-dose) on single dose; Hour 0(pre-dose) of day1, day8, day15, day28 on multiple dose of first cycle; hour 0(pre-dose) of day15, day28 of second and third cycle; hour 0(pre-dose) of day28 of fourth to eighth cycle.Each cycle is 28 days.
  Correlation between 2-hydroxyglutaric acid and efficacy

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The Affiliated Hosptial of Xuzhou Medical University, Xuzhou, Jiangsu
  - Tianjing Medical University Cancer Institute&Hospital, Tianjin, Tianjin Municipality
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hosptial Zhejiang University School of Medical, Hangzhou, Zhejiang